CLINICAL TRIAL: NCT07145658
Title: A Randomised Placebo-controlled Trial Assessing the Effect of Daily Supplementation of a 20-ingrediant Multivitamin, on Markers of Health, Wellbeing and Cognitive Function in Healthy Volunteers
Brief Title: Multivitamin for Health and Cognition
Acronym: Vitals+
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Anthony Hobson (Other)
Collaborators: Heights (Industry)
Responsible Party: Sponsor-Investigator, Dr Anthony Hobson, Clinical Director, The Functional Gut Clinic
Organization: The Functional Gut Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: FGC-25-01
Record Dates: First submitted 2025-08-05; First posted 2025-08-28 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-08

CONDITIONS: Healthy; Cognition; Health
Keywords: multivitamin
MeSH Terms: interventions — Geritol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): 90 days placebo capsules 2x daily
  Interventions: Dietary Supplement: Placebo Capsule(s)
- Multivitamin (Experimental): 90 days multivitamin capsules 2x daily
  Interventions: Dietary Supplement: multivitamin

INTERVENTIONS:
Dietary Supplement: Placebo Capsule(s) — Placebo - identical capsules containing inert colour matched power
  Arms: Placebo
Dietary Supplement: multivitamin — 20-ingredient multivitamin
  Arms: Multivitamin

SUMMARY:
Multiple factors contribute to poor mental and cognitive health including well-balanced nutrition. This research project will aim to establish whether a the multivitamin Vitals+ is more effective in improving markers of health, well being and cognitive function, in healthy volunteers compared to placebo.

The study aims to recruit 36 healthy volunteers for a placebo controlled double blind design. Participants will be screened through a phone call to ensure they meet the appropriate inclusion and exclusion criteria to enter the study before attending the clinic for tests to assess blood based vitamin and minerals levels, cognitive function, well-being questionnaires and tests to look at function of their gut barrier and activity of gut bacteria. They will then take the multi-vitamin or a placebo daily for 3 months before repeating the same tests in a second in person clinic appointment.

ELIGIBILITY:
Inclusion Criteria:

1. Participant has provided written informed consent before participating in the study after being given a full description of the study and prior to any study-specific procedures being performed.
2. Participant has no significant medical diagnosis (health individuals)
3. Participant takes no regular prescription medication
4. Participant is not undertaking any restrictive diet (e.g. Carnivore, Low FODMAP)
5. Participant agrees to adhere to guidance on fortified food intake for the duration of the study
6. Participant is a male or non-pregnant female and is 18-70 years of age
7. If WOCBP participant is willing to adhere to one of the following methods of contraception i) Hormonal contraception e.g. the 'pill' or an implant ii) Intrauterine device (IUD) iii) Intrauterine hormone-releasing system (IUS) iv) Hysterectomy v) Vasectomised partner vi) Sexual abstinence (if it is in line with your preferred and usual lifestyle).
8. Participant can communicate well with the Investigator and to comply with the requirements for the entire study.
9. Participant has capacity to understand written English.
10. Participant has a body mass index (BMI) of 18.5 - 39.9kg/m2 (bounds included).
11. Participant agrees to follow all pre-test preparation before L/M-HMBT testing.

Exclusion Criteria:

1. Participant has consumed nutritional supplement in the past 3 months
2. Diagnosis of any current medical condition, except visual impairment and other conditions at the discretion of the investigator
3. Participated in a trial of an investigational medical product or medical device in the last 28 days.
4. Females who report to be pregnant or lactating
5. Prior abdominal surgery
6. Unwilling to maintain a stable diet for the duration of the trial.
7. Unable to comply with limiting fortified food intake to <5 portions per week for the duration of the study
8. Being in the opinion of the investigator unsuitable
9. Insufficient knowledge of English to complete the daily bowel diary and food diary.
10. Hypersensitivity to any component of the supplement
11. Hypersensitivity or known allergy to lactulose or mannitol.
12. Consumption of oral antibiotics in the last 4 weeks.
13. NSAIDs for 2 weeks prior to and during the entire 90 day study period. Participant should not be a chronic NSAID user (>1 day/week).
14. Gastrointestinal infection in the past 4 weeks.
15. IV vitamin/mineral therapy in the past 12 weeks
16. Use of medical devices for the purpose of cognitive enhancement, such as neural stimulation, in the 2 weeks prior or during the study period
17. Participant is involved in this study as an Investigator, sub-Investigator, study coordinator, other study staff, or Sponsor member.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-07-07 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Cognitive function score | Start of study to end of study (3 months)
  Mean change in cognition function score from start of study to end of study between multivitamin and placebo groups.
  Cognitive function test - a validated, self-administered tool providing a composite score combining subscores of executive function, processing speed, episodic memory, recognition memory and overall dementia risk index. A higher score indicates better cognitive function.

SECONDARY OUTCOMES:
Product safety | start of study to end of study (3 months)
  Product safety assessed by number of adverse events raised by clinically significant changes in standard haematology and biochemistry panels in the active group.
Mean change in The Profile of Mood States questionnaire (POMS) | Start of study to end of study (3 months)
  The Profile of Mood States questionnaire (POMS), is a validated psychological test that contains 65 words and statements that describe feelings. The questionnaire is used to assess changes in mood states overtime, including: Tension, Anger, Fatigue, Depression, Confusion and Vigour. For each word or statement a 5 point Likert scale is utilised to describe the most applicable answer to the word or statement. A total mood disturbance score can be calculated based on the responses.
Mean change in GHQ-12 | start of study to end of study (3 months)
  The General Health Questionnaire-12 (GHQ-12) is a 12-question survey that screens for mental health problems. It is a short version of the original 60-item General Health Questionnaire (GHQ). The questionnaire is often used in the primary care setting and includes questions relating to sleep, tension, temperament, and social functioning difficulties. Each question is measured on a 4 point Likert scale.
Serum B12 | start of study to end of study (3 months)
  Comparison of mean change in levels of serum B12 (pg/ml) from start of study to end of study, between active and placebo groups
Homocysteine | start of study to end of study (3 months)
  Comparison of mean change in levels of Homocysteine (umol/L) from start of study to end of study, between active and placebo groups
Vitamin B6 | start of study to end of study (3 months)
  Comparison of mean change in levels of Plasma PLP (Vitamin B6)(ug/L) from start of study to end of study, between active and placebo groups
Vitamin D | start of study to end of study (3 months)
  Comparison of mean change in levels of Vitamin D(pmol/L) from start of study to end of study, between active and placebo groups
HbA1c | start of study to end of study (3 months)
  Comparison of mean change in levels of HbA1c (%) from start of study to end of study, between active and placebo groups
Iron | start of study to end of study (3 months)
  Comparison of mean change in levels of Iron (umol/L) from start of study to end of study, between active and placebo groups
Riboflavin (Vitamin B2) | Start of study to end of study (3 months)
  Comparison of mean change in levels of Riboflavin (vitamin B2) between active and placebo groups, measured using Erythrocyte glutathione reductase activation coefficient (EGRAC) with a higher value indicating lower riboflavin levels

OTHER OUTCOMES:
Changes in Intestinal permeability | start of study to end of study (3 months)
  Two sugars (lactulose/mannitol) are ingested at a controlled amount with ratio in urine samples provided over 3 hours measured to determine gut/barrier dysfunction
Correlation between HMBT results and changes in blood-based biomarkers | start of study to end of study (3 months)
  Lactulose Hydrogen Methane Breath Testing (HMBT) is a test utilised clinically to diagnose both Small Intestinal Bacterial Overgrowth (SIBO) and Intestinal Methanogenic Overgrowth (IMO). Total production of hydrogen and methane (area under curve) will also be assessed using this method.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - The functional gut clinic, London
  - The functional gut clinic, Manchester

IPD SHARING:
Plan to Share IPD: No